CLINICAL TRIAL: NCT03776851
Title: Effect of Erythropoietin on Red Blood Cell Requirement in Children With Hemolytic Uremic Syndrome: a Randomized Controlled Trial
Brief Title: Erythropoietin in Hemolytic Uremic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Principal Investigator, Alejandro Balestracci, Principal Investigator, Hospital General de Niños Pedro de Elizalde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 347-HGNPE-2018
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Hemolytic-Uremic Syndrome; Anemia
Keywords: Hemolytic-Uremic Syndrome; erythropoietin; RBC transfusion
MeSH Terms: conditions — Hemolytic-Uremic Syndrome; Anemia | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythropoietin (Experimental): Erythropoietin plus standard of care (RBC transfusions if Hb ≤7 mg/dl and/or hemodynamic instability)
  Interventions: Drug: erythropoietin
- No Intervention (No Intervention): Standard of care: RBC transfusions if Hb ≤7 mg/dl and/or hemodynamic instability

INTERVENTIONS:
Drug: erythropoietin — erythropoietin 50 International Units (IU) per kilogram three times weekly by subcutaneous route
  Other Names: EPO
  Arms: Erythropoietin

SUMMARY:
This study will evaluate the impact of early administration of erythropoietin in the number of red blood cell transfusions in children with Shiga toxin-producing Escherichia coli hemolytic uremic syndrome (STEC-HUS).

DETAILED DESCRIPTION:
Introduction:

Anemia in STEC-HUS is treated with red blood cell (RBC) transfusions. It can causes hypervolemia, hyperkalemia, exacerbate the thrombotic state of the disease, transmit infectious agents and trigger antigenic sensitization. Anemia is mainly due to hemolysis, but deficit of erythropoietin synthesis (EPO) may aggravate it. Although recombinant human EPO is frequently used in children with STEC-HUS there is no adequate evidence of its benefit. If it is confirmed that EPO reduce the number of RBC transfusions, its administration could diminish the aforementioned risks and also reduce costs.

Objective:

To determine if EPO administration decreases the number of RBC transfusions and; secondarily, to assess if its levels influence on transfusion requirement.

Methodology:

Randomized, open controlled clinical trial. We will include 28 patients (14 per arm) <18 years with STEC-HUS admitted to our hospital. They will be grouped after randomization:(1) One to standard of care (RBC transfusions with hemoglobin ≤7 mg / dl and/or hemodynamic instability) and (2) the other to standard of care plus EPO (50 u / kg subcutaneous three times weekly) and RBC transfusions with hemoglobin ≤7 mg / dl). Serum EPO will be measured by ELISA and together with the clinical and laboratory variables, association with RBC transfusions number will be sought. Written informed consent and assent when appropriate, will be requested prior to enter into the study.

ELIGIBILITY:
Inclusion Criteria:

* Post diarrheal HUS: Prodrome of enteritis followed by microangiopathic hemolytic anemia, thrombocytopenia and signs of renal damage (increased plasma creatinine, proteinuria, and / or hematuria). Proven STEC infection wiil not be required to enter into the study.

Exclusion Criteria:

* Atypical HUS
* HUS associated with systemic diseases (pneumococcal infection, HIV, Systemic lupus erythematosus) or drugs
* Anemia or known kidney disease
* Previously transfused or treated with erythropoietin
* Contraindications to erythropoietin

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of RBC transfusions | At the end of the 36 month study recruiting period
  To determine if administration of erythropoietin decreases the number of RBC during the acute stage of hemolytic uremic syndrome

SECONDARY OUTCOMES:
Erythropoietin levels | At the end of the 36 month study recruiting period
  To determine if erythropoietin levels correlate with RBC transfusions requirement.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Balestracci, MD, PhD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- HGNPE, CABA, Argentina

IPD SHARING:
Plan to Share IPD: Yes
The authors will share the generated data with qualified external researchers during the next 5 years after article publication. All data provided will be anonymized to respect the privacy of patients who have participated in the trail in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: During the next 5 years after article publication.
Access Criteria: Qualified external researchers

REFERENCES:
- [Background] Ardissino G, Dacco V, Testa S, Civitillo CF, Tel F, Possenti I, Belingheri M, Castorina P, Bolsa-Ghiringhelli N, Tedeschi S, Paglialonga F, Salardi S, Consonni D, Zoia E, Salice P, Chidini G. Hemoconcentration: a major risk factor for neurological involvement in hemolytic uremic syndrome. Pediatr Nephrol. 2015 Feb;30(2):345-52. doi: 10.1007/s00467-014-2918-0. Epub 2014 Aug 23. PMID 25149851
- [Background] Scheiring J, Rosales A, Zimmerhackl LB. Clinical practice. Today's understanding of the haemolytic uraemic syndrome. Eur J Pediatr. 2010 Jan;169(1):7-13. doi: 10.1007/s00431-009-1039-4. Epub 2009 Aug 26. PMID 19707787
- [Background] Exeni R, Donato H, Rendo P, Antonuccio M, Rapetti MC, Grimoldi I, Exeni A, de Galvagni A, Trepacka E, Amore A. Low levels of serum erythropoietin in children with endemic hemolytic uremic syndrome. Pediatr Nephrol. 1998 Apr;12(3):226-30. doi: 10.1007/s004670050443. PMID 9630043
- [Background] Moore E, Bellomo R. Erythropoietin (EPO) in acute kidney injury. Ann Intensive Care. 2011 Mar 21;1(1):3. doi: 10.1186/2110-5820-1-3. PMID 21906325
- [Background] Warady BA, Silverstein DM. Management of anemia with erythropoietic-stimulating agents in children with chronic kidney disease. Pediatr Nephrol. 2014 Sep;29(9):1493-505. doi: 10.1007/s00467-013-2557-x. Epub 2013 Sep 5. PMID 24005791
- [Background] Pape L, Ahlenstiel T, Kreuzer M, Drube J, Froede K, Franke D, Ehrich JH, Haubitz M. Early erythropoietin reduced the need for red blood cell transfusion in childhood hemolytic uremic syndrome: a randomized prospective pilot trial. Pediatr Nephrol. 2009 May;24(5):1061-4. doi: 10.1007/s00467-008-1087-4. Epub 2008 Dec 16. PMID 19085014
- [Background] Balestracci A, Martin SM, Toledo I, Alvarado C, Wainsztein RE. Early erythropoietin in post-diarrheal hemolytic uremic syndrome: a case-control study. Pediatr Nephrol. 2015 Feb;30(2):339-44. doi: 10.1007/s00467-014-2911-7. Epub 2014 Aug 21. PMID 25138373
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879
- [Derived] Balestracci A, Capone MA, Meni Battaglia L, Toledo I, Martin SM, Beaudoin L, Balbaryski J, Gomez L. Erythropoietin in children with hemolytic uremic syndrome: a pilot randomized controlled trial. Pediatr Nephrol. 2022 Oct;37(10):2383-2392. doi: 10.1007/s00467-022-05474-9. Epub 2022 Feb 15. PMID 35166922